CLINICAL TRIAL: NCT02221258
Title: Phase 1 Clinical Trial to Evaluate the Safety of FURESTEM-RA Inj. in Patients With Moderate to Severe Rheumatoid Arthritis
Brief Title: Safety of FURESTEM-RA Inj. in Patients With Moderate to Severe Rheumatoid Arthritis(RA)
Acronym: RA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kang Stem Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSB-RA
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2015-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Rheumatic Disease; RA; Stem cell; Cell therapy; furestem; Umbilical cord Blood; hUCB-MSC; UCB-MSC
MeSH Terms: conditions — Arthritis, Rheumatoid; Rheumatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FURESTEM-RA Inj.+DMARDs (Experimental): FURESTEM-RA Inj. 1. 2.5x10^7 stem cells+DMARDs after registration FURESTEM-RA Inj. 2. 5.0x10^7 stem cells+DMARDs after registration FURESTEM-RA Inj. 3. 1.0x10^8 stem cells+DMARDs after registration
  Interventions: Biological: FURESTEM-RA Inj.

INTERVENTIONS:
Biological: FURESTEM-RA Inj. — Patients will be treated FURESTEM-RA Inj.+DMARDs(Disease-Modifying antirheumatic drugs)

SUMMARY:
The purpose of phase 1 clinical trial is to to evaluate safety in subjects with moderate to severe rheumatoid arthritis after infusion.

DETAILED DESCRIPTION:
Rheumatoid arthritis(RA) is a chronic and progressive autoimmune disease characterized by synovial hyperplasia and joint damage leading to clinically significant functional impairment. In RA, for some unknown reason, immune cells infiltrate into synovium of joint and produce the 'rheumatoid factor', prostaglandins, cytokines and other mediators. It damages joint and cartilage, even other organs. 80% of the RA patients have Rheumatoid factor which is caused by high expression ratio of auto-antibodies in blood. Produced immune complexes, immune cells and antigen-presenting cells(including macrophages, B cells, dendritic cells) activate and release cytokines and then synovial tissue becomes thickened and damaged.

It has been reported that synthetic DMARDs(disease-modifying antirheumatic drugs) including methotrexate(MTX), sulfasalazine and biological DMARDs such as tumor necrosis factors(TNF)-α blockers, abatacept and rituximab, often in combination with MTX, are effective. But they still are limited by lack or loss of efficacy in certain patients and serious complications such as serious infections and malignancies. So, there is a need to identify new treatment.

FURESTEM-RA Inj. is composed of allogeneic hUCB-MSC(human Umbilical Cord Blood derived-Mesenchymal Stem cell). hUCB-MSCs are mesenchymal stem cells from umbilical cord blood. Mesenchymal stem cells are well-known for immunosuppression, anti-inflammatory ability and capable of differentiating into a wide range of cell types including osteocytes and chondrocytes. Therefore, FURESTEM-RA Inj. has huge possibility as cell therapy products for RA patients.

ELIGIBILITY:
Inclusion Criteria:

1. of either gender, 19-80years old
2. Subjects must be diagnosed with ACR functional class I. II, III Rheumatoid Arthritis according to the 2010 ACR/EULAR criteria for at least 12 weeks duration.
3. Subjects must be taking DMARDs or NSAIDs including methotrexate, sulfasalazine, hydroxychloroquine, leflunomide of stable dose within 12 weeks before screening visit and be willing to remain on stable dose throughout the study
4. If subject is currently administering steroids everyday, when steroid dose is converted into prednisolone oral dose, the subject should take a stable dose(≤10mg/day) over 4 weeks on screening visit
5. Subject who has moderate to severe disease activity (DAS28-ESR>3.2) on screening visit
6. Subject who understands and voluntarily sign an informed consent form

Exclusion Criteria:

1. Subjects who is diagnosed ACR function class IV Rheumatoid Arthritis
2. Subjects who has cardiovascular disorders, blood dyscrasia, AIDS(Acquired Immune Deficiency Syndrome), other rheumatic disease(Crohn's disease, systemic lupus erythematosus, lyme disease, psoriatic arthritis, spondylarthropathy, infectious or reactive arthritis, reiter's syndrome, etc.)
3. subject who has administered the following biological DMARDs

   * subject who has administered more than 1 drugs(Infliximab, Adalimumab, Etanercept, Anakinra, Abatacept) within 6 months before screening visit
   * subject who has administered Rituximab within 1 year before screening visit
4. Subject who has history of hypersensitivity, heavy metal poisoning, etc. to drugs which is composed of similar components.
5. Subject who has treated intra-articular steroid injection within 4 weeks before screening visit
6. Subject who has administered ACTH(adrenocorticotropic hormone) agents within 4 weeks before screening visit
7. Subject who has undergone administration of any investigational drug within 30 days before screening visit.
8. Subject who has diseases or takes medicine which are prohibited prescription of NSAIDs.
9. Subject who needs to take the medicine which is prohibited to take at the same time
10. Pregnant, breast-feeding women
11. Subject who has sever dyshepatia (Serum creatinine level ≥ 1.7mg/dl)
12. Subject who has severe renal dysfunction (ALT/AST/bilirubin value ≥ 2 upper limit of the normal range at screening test)
13. Any other condition which the PI Judges would make patient unsuitable for study participation
14. Subject who experienced stem cell therapy

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Safety of FURESTEM-RA Inj. treatment | 4 weeks follow-up after treatment
  Evaluate the number of adverse events, including clinically significant changes in physical examination, safety lab tests, ECG, vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Kichul Shin, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul national University Boramae medical center, Seoul, Seoul, South Korea